CLINICAL TRIAL: NCT00319540
Title: A Randomized Controlled Trial of a Psychoeducational Group Program for Unipolar Depression in Adults in Norway
Brief Title: RCT of Psychoeducational Program of Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2906
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2001-01

CONDITIONS: Unipolar Depression
Keywords: Depression; psychoeducation; RCT; primary health services
MeSH Terms: conditions — Depressive Disorder; Depression

INTERVENTIONS:
Behavioral: Control with depression course (CWD)

SUMMARY:
The purpose of the study is to test the efficacy of a psychoeducational group program on unipolar depression

DETAILED DESCRIPTION:
Unipolar depression is a common disorder which may be treated by drugs or psychological intervention. Many patients prefer psychological treatment, but there is a lack of professional skills and methods for effectively dealing with this in the primary health services,where most of the depressed patients are seen.For this reason it is of great importance to develop and test psychological methods which may be applied in the primary health services, as well as in the specialized psychiatric services.In the present study a psychoeducational group method is tested, with trained psychiatric nurses as the most common group leaders.

Comparison: People with unipolar depression receiving "treatment as usual"

ELIGIBILITY:
Inclusion Criteria:Unipolar depression -

Exclusion Criteria:Psychosis, other psychiatric disorders, subclinical depression, suicidal ideation, learning disabilities

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155
Dates: Start 2001-03; Study Completion 2002-03

PRIMARY OUTCOMES:
BeckDepression Inventory : A questionnaire with 23 items to measure symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: Odd Steffen Dalgard, M.D., Ph.D., Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

REFERENCES:
- [Derived] Ducasse D, Courtet P, Seneque M, Genty C, Picot MC, Schwan R, Olie E. Effectiveness of the first French psychoeducational program on unipolar depression: study protocol for a randomized controlled trial. BMC Psychiatry. 2015 Nov 17;15:294. doi: 10.1186/s12888-015-0667-7. PMID 26578205